CLINICAL TRIAL: NCT05771623
Title: Botulinum Toxin Type a Iontophoresis for Postburn Hypertrophic Scar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hayam Mahmoud Aboulmaati Alnawagy, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003749
Record Dates: First submitted 2023-02-14; First posted 2023-03-16 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Hypertrophic Scar
Keywords: Hypertrophic scar
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Control group: (38 patients with hypertrophic scar) receive traditional PT for postburn scar.
  Study group: (38 patients with hypertrophic scar) receive botulinum toxin type a iontophoresis plus traditional PT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum Toxin Type a Iontophoresis for Postburn Hypertrophic Scar (Experimental): The study group includes 38 postburn hypertrophic scar patients l receiving Botox iontophoresis once monthly for 3 months; in addition to their physical therapy program (Stretching exercises, Pressure Therapy and Massage) 2 sessions per week for 3 months.
  Botulinum toxin type A (Botox Allergan ®, Irvine, CA, USA) is used. 100 U vacuum-dried powder in a single-use vial for reconstitution diluted in 2 mL of sterile, preservative-free 0.9% saline to constitute a solution at a concentration of 4 U/0.1 mL) is being administered once a month for a total period of three months.
  The dose will be adjusted to 2.5 U/cm2 of the scar. The dose shouldn't exceed 100 units per session.
  Interventions: Device: Iontophoresis drug delivery device; Behavioral: Traditional physical therapy
- Traditional physical therapy for postburn hypertrophic scar (Active Comparator): This group includes 38 patients with postburn hypertrophic scar who will receive the traditional PT (deep friction massage, stretching and pressure therapy).
  Interventions: Behavioral: Traditional physical therapy

INTERVENTIONS:
Device: Iontophoresis drug delivery device — Botulinum toxin type A (Botox Allergan ®, Irvine, CA, USA) is used. 100 U vacuum-dried powder in a single-use vial for reconstitution diluted in 2mL of sterile, preservative-free 0.9% saline to constitute a solution at a concentration of 4 U/0.1 mL) is being administered once a month for a total period of three months.
  The dose will be adjusted to 2.5 U/cm2 of the scar. The dose shouldn't exceed 100 units per session.
  This can be done through the Iontophoresis drug delivery device. Traditional PT: Stretching, deep friction massage and pressure therapy (2 times per week for 3 months).
  Arms: Botulinum Toxin Type a Iontophoresis for Postburn Hypertrophic Scar
Behavioral: Traditional physical therapy — Traditional PT: Stretching, deep friction massage and pressure therapy (2 times per week for 3 months).

SUMMARY:
The goal of this clinical trial study: is to determine the effect Botulinum toxin type A iontophoresis in hypertrophic scars for post burned patients. The main question is it aims to answer is:

* Does Botulinum toxin type A iontophoresis may help in minimizing postburn hypertrophic scars?
* Participants will receive the treatment for 3 months.
* Assessment will be done before and after treatment.

DETAILED DESCRIPTION:
1. Subjects:

   Seventy-six Patients from both genders who have post burn hypertrophic scar will participate in this study. Their ages will be ranged 20 to 40 years.
2. Design of the study:

In this study the patients will be randomly assigned into two equal groups (38 patients for each group):

1. Group A (Study group):

   This group includes 38 patients who will receive botulinum toxin type A iontophoresis once monthly for 3 months, in additional to traditional physical therapy (Positioning, Stretching exercises, Pressure Therapy and Massage) 2 sessions per week for 3 months.
2. Group B (Control group):

   This group includes 38 patients who will receive traditional physical therapy (Positioning, Stretching exercises, Pressure Therapy and Massage) 2 sessions per week for 3 months.

   - Equipments:

   Measurement equipments:
   1. Sonography:

      It is high-resolution B-image sonogram which allows a good penetration depth of up to 40 mm into the skin and a resolution of around 158 micro m. It has been successfully utilized for objectively measuring pathological scars.
   2. Patient and Observer Scar Assessment Scale (POSAS):

      It consists of two parts; one for the patient (Patient scale; POSAS Patient) and one for the physician (Observer scale; POSAS Observer). Both contain six items on a 10-point rating scale and an extra category "Overall Opinion". All characteristic features of the pathological scars are covered by the questionnaire: vascularity, pigmentation disorders, relief/texture, thickness, pliability, surface area, pain, and itching/pruritus. The latter items, in particular, concern the well-being of the patients.
      * Sonography:

        • High frequency ultrasound is the most common used technique for scar assessment.

        • The working mechanism is based on refection of sound waves of structures with different acoustic impedances and the analysis of the refection time to determine the depth of the structure.

        • The penetration depth ranges from the upper dermal layers to full-thickness skin and subcutaneous structures, depending on the employed frequency b. Patient and Observer scar Assessment Scale (POSAS):

        • The scar will be rated numerically on a ten-step scale by both the patient and doctor.

        • Six items on the Observer Scale: vascularity, pigmentation, thickness, relief, pliability, and surface area.

        • The Patient Scale consists of pain, itchiness, color, stiffness, thickness, and irregularity of the scar.
        * One of the reasons POSAS was chosen for scar evaluation is because it is the only scar assessment tool to include a component for patients to fill in.
        * Furthermore, its distinctive feature of reflecting subjective symptoms like pain and pruritus and because of its appropriateness for everyday practice.
        * Both sonography and POSAS will be used for assessment of hypertrophic scar pre-treatment and post treatment (after 3 months then after 6 months as follow up).
      * Procedures of iontophoresis drug delivery device:

      the iontophoresis group will receive botulinum toxin type A iontophoresis using an iontophoretic drug delivery system (Phoresor IIAuto,Model PM850, IOMED.) - Procedures of botulinum toxin type A iontophoresis:

      • Botulinum toxin type A (Botox Allergan ®, Irvine, CA, USA) will be used.

      • 100 U vacuum-dried powder in a single-use vial for reconstitution diluted in 2 mL of sterile, preservative-free 0.9% saline to constitute a solution at a concentration of 4 U/0.1 mL) will be administered once a month for a total period of three months.
      * The dose will be adjusted to 2.5 U/cm2 of the lesion.
      * The dose shouldn't exceed 100 units per session.

        * Physical therapy program for both groups:

      traditional physical therapy (Positioning, Stretching exercises, Pressure Therapy and Massage) 2 sessions per week for 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patient with hypertrophic scar (3-6) months after burn healing.
* Age range between 20-40 years.
* Male and female patients will participate in the study.
* All patients have a postburn hypertrophic scar at different body sites.
* All patients enrolled on the study will have their informed consent.

Exclusion Criteria:

* Patients with prior medical histories of cardiac arrhythmias.
* Patients with cardiac pacemakers.
* Patients with orthopedic implants.
* Areas of skin with lesions and impaired sensation.
* During pregnancy and breastfeeding.
* Patient with diabetes mellitus.
* Patients with a history of hypersensitivity or adverse reactions associated with (BTX_A).
* Recent BTA administration 6 months before the study.
* Any subject complaining of psychiatric disorders or neurological disorders such as myasthenia gravis.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
High resoluton ultrasonography | Change of hypertrophic scar thickness from the beginning of treatment to the end of treatment(after 3 months from the beginning of treatment).
  High frequency ultrasound is the most common used technique for scar assessment. Its inferior resolution compared to optical equivalents is mitigated by its superior penetration depth allowing thickness analysis, even in severe scar thickening. The working mechanism is based on refection of sound waves of structures with different acoustic impedances and the analysis of the refection time to determine the depth of the structure. The penetration depth ranges from the upper dermal layers to full-thickness skin and subcutaneous structures, depending on the employed frequency.
Patient and observer scar assessment scale | Assessing the change of patient and observer scar assessment scale score from baseline (beginning of treatment) to 3 months after treatment.
  The scar will be rated numerically on a ten-step scale by both the patient and doctor on six items: vascularity, pigmentation, thickness, relief, pliability, and surface area on the Observer Scale. The Patient Scale consists of pain, itchiness, color, stiffness, thickness, and irregularity of the scar. Minimal score means good progression and maximum score means the scare is worse.

OTHER OUTCOMES:
High resoluton ultrasonography | Change of hypertrophic scar thickness from the beginning of treatment to 6 months after treatment.
  High frequency ultrasound is the most common used technique for scar assessment. Its inferior resolution compared to optical equivalents is mitigated by its superior penetration depth allowing thickness analysis, even in severe scar thickening. The working mechanism is based on refection of sound waves of structures with different acoustic impedances and the analysis of the refection time to determine the depth of the structure. The penetration depth ranges from the upper dermal layers to full-thickness skin and subcutaneous structures, depending on the employed frequency.
Patient and observer scar assessment scale | Assessing the change of patient and observer scar assessment scale score from baseline (beginning of treatment) to 6 months after treatment.
  The scar will be rated numerically on a ten-step scale by both the patient and doctor on six items: vascularity, pigmentation, thickness, relief, pliability, and surface area on the Observer Scale. The Patient Scale consists of pain, itchiness, color, stiffness, thickness, and irregularity of the scar. Minimal score means good progression and maximum score means the scare is worse.

CONTACTS AND LOCATIONS:
Overall Officials: A M Abd Elbaky, Professor, Study Director — faculty of physical therapy
Locations (1):
- Faculty of physical therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT05771623/Prot_SAP_000.pdf